CLINICAL TRIAL: NCT05713682
Title: Prevalence of Peri-implantitis Between Periodontitis and Nonperiodontitis Sites Treated With Alveolar Ridge Preservation: A Retrospective Cohort Study
Brief Title: Peri-implantitis Between Periodontitis and Nonperiodontitis Sites With ARP
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20200275
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis, periodontitis, alveolar ridge preservation
MeSH Terms: conditions — Peri-Implantitis; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: alveolar ridge preservation — bone grafting at extracted sites

SUMMARY:
The goal of this observational study is to compare the prevalence of peri-implantitis between periodontitis and nonperiodontitis sites treated with alveolar ridge preservation.

The main question it aims to answer is:

• whether the occurrence of PI is associated with reasons for dental extraction because of periodontitis and nonperiodontitis after alveolar ridge preservation.

Researchers will compare the prevalence of peri-implantitis between periodontitis and nonperiodontitis sites treated with alveolar ridge preservation.

ELIGIBILITY:
Inclusion Criteria

1. patients aged ≥ 20 years
2. patients who required tooth extraction and implant therapy
3. at least two bite-wing radiographs: baseline and at least a 6-month follow-up

Exclusion Criteria

1. a medical condition as a contraindication to dental surgery, autoimmune disorder, immunosuppression, or uncontrolled diabetes (HbA1c > 7%);
2. ong-term nonsteroidal anti-inflammatory drug use
3. oral bisphosphonate therapy
4. pregnancy or lactation
5. the absence of follow-up bite-wing radiograph
6. cigarette consumption >10 per day
7. a history of head and neck radiotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled consecutive patients who received dental extraction and ARP simultaneously and dental implant treatment at least 4 months after ARP at the Division of Periodontics, Kaohsiung Medical University Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
occurrence of peri-implantitis | 2013-2020
  bone loss at implant sites

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Chou, Master, Study Chair — School of Dentistry, College of Dental Medicine, Kaohsiung Medical University, Kaohsiung, Taiwan